CLINICAL TRIAL: NCT03319602
Title: Effect of a Double Trunk Mask Associated to Nasal Prongs During a High Flow Oxygenation Method
Brief Title: Effect of a Modified Oxygen Mask Associated to Nasal Prongs During a High Flow Oxygenation Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratory of Movement, Condorcet, Tournai, Belgium (Other)
Responsible Party: Principal Investigator, frédéric Duprez, Research collaborator, Laboratory of Movement, Condorcet, Tournai, Belgium
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HFODTM01
Record Dates: First submitted 2017-10-05; First posted 2017-10-24 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Oxygen Inhalation Therapy
Keywords: oxygen mask; high-flow oxygen therapy; acute respiratory failure

STUDY DESIGN:
Intervention Model Description: Comparison of level oxygenation between classical oxygenation with nasal canulae with or without adjunctive of a double trunk mask
Who Masked: Outcomes Assessor
Masking Description: Assessor blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygenation only with nasal canula (Active Comparator): intervention: classical oxygenation with nasal canula (High flow)
  Interventions: Device: Double trunk mask add above a nasal canulae
- Oxygenation with double trunk masknasal canula (Experimental): oxygenationwith DTM above nasal canula
  Interventions: Device: Double trunk mask add above a nasal canulae

INTERVENTIONS:
Device: Double trunk mask add above a nasal canulae — oxygenation only with nostril prongs

SUMMARY:
The aim of this study is to determine the effect (on PaO2) of a modified mask associated to nasal cannula used for high flow oxygenation.

DETAILED DESCRIPTION:
Study Design This is a single-center, randomized, blind investigator, 2-way crossover study design. Enrolled participants had severe hypoxia being treated at Intensive Care Unit associated with a hospital in Hornu (Epicura).

The study consisted of two intervention periods of 2 weeks separated by a washout period of 20 minutes. (Figure 1) The objective of the study is to determine whether adjunctive mask of our design (Double Trunk Mask - DTM) has an effect on increasing arterial pressure in Oxygen (PaO2) diagnosed with severe hypoxia.

The protocol and informed consent documents were reviewed and approved by a recognized ethics review board at the study facility. The study was performed in accordance with the Declaration of Helsinki.

Statistical Analysis

All participants who received this intervention and completed two phases of study were included in the efficacy analysis.

A sample size of 15 participants was needed to provide 90% power to detect a 10 mm Hg difference in PaO2. ANOVA for repeated measures followed by a post hoc test were used to compare the difference between participants receiving (CHFONP + DTM) and CHFONP alone.

The test was performed with a significance level of 0.05 (two-sided). Statistical analyses were carried out using SigmaPlot software version 11.0 (Systat Software Inc. UK).

Adverse Event Assessment

Safety was assessed by the number of participants with adverse events (AEs). AEs were collected by systematic assessment using terms from the Medical Dictionary for Regulatory Activities (MedDRA), version 11.1 in participants who received one or more doses of intervention. Adverse events during washout were not collected.

ELIGIBILITY:
Inclusion Criteria:

Regardless of gender, at least 18 years of age and diagnosed with severe Hypoxia (PaO2/FiO2 < 300 mm Hg), dyspnea with severe rest at stake accessory muscles of respiration, respiratory rate (RR) ≥ 25 CPM, PaCO2 ≤ 45 mmHg, patient with an arterial catheter and without hemodynamic instability, Glasgow Coma Scale ≥ 12/15, written consent. Participants were also required to have a sufficient level of education to understand study procedures and be able to communicate with site personnel.

Exclusion Criteria Patients were excluded if they Hypercapnia (> 45 mm Hg with respiratory acidosis), cardiogenic pulmonary edema, COPD, pulmonary fibrosis, hypoventilation obesity syndrom, arterial pressure < 60 mm Hg or treatment by epinephrine > to 0,1 gamma/kg/minute, deterioration of awareness (Glasgow scale < or = 12), acute confusional state.

Participants were randomized in a 1:1 ratio to receive either (CHFONP) classical High Flow Oxygenation with nasal prongs (20 minutes) or CHFNOP with an adjunctive of a DTM.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-09-02 (Actual)

PRIMARY OUTCOMES:
Level of blood oxygenation (PaO2) after adjunction of a double trunk mask to a high flow oxygen canulae | 4 hours
  The primary endpoint was the change of PaO2. Sequence (Figure 1): The patient should be placed in semi-seated (position at 45 °) Patient will be oxygenated with high-fow nasal cannula (HFNC). Fraction delivered in Oxygen and flow rate will be adjusted to obtain a Saturation in oxygen > at 90%.
  1. Arterial gazometry will be taken after 20 and 60 minutes wih HFNC.
  2. The clinician will associate the Double Trunk Mask (DTM) with the same parameters of the high-fow nasal cannula. Arterial gazometry will be performed after 20 and 60 minutes after placement of DTM.
  3. After the withdrawal of DTM, arterial gazometry will be performed after 20 and 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: frédéric mr duprez, Msc, Principal Investigator — Condorcet
Locations (1):
- epicura Hornu, Hornu, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hnatiuk OW, Moores LK, Thompson JC, Jones MD. Delivery of high concentrations of inspired oxygen via Tusk mask. Crit Care Med. 1998 Jun;26(6):1032-5. doi: 10.1097/00003246-199806000-00022. PMID 9635651
- [Result] Chechani V, Scott G, Burnham B, Knight L. Modification of an aerosol mask to provide high concentrations of oxygen in the inspired air. Comparison to a nonrebreathing mask. Chest. 1991 Dec;100(6):1582-5. doi: 10.1378/chest.100.6.1582. PMID 1959399

DOCUMENTS (2):
  • Informed Consent Form (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT03319602/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT03319602/Prot_SAP_002.pdf